CLINICAL TRIAL: NCT01337076
Title: Evaluation of a Revised Indication for Determining Adult Cochlear Implant Candidacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM-EXP-A2010-01
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cochlear implant (Other)
  Interventions: Device: cochlear implant

INTERVENTIONS:
Device: cochlear implant — Cochlear implant surgery
  Other Names: implantable hearing device

SUMMARY:
The Sponsor values the progression of hearing healthcare practice and acknowledges a need for re-evaluation of indications for determining adult cochlear implant candidacy. This need arises from current research, peer reviewed literature, and technological advancement with concomitant performance outcomes. To address this specifically, the Sponsor proposes to evaluate the safety and efficacy of the Cochlear™ Nucleus® implant system with a revised indication.

DETAILED DESCRIPTION:
Existing research, as discussed, supports the opinion that current candidacy criteria are set conservatively. The Sponsor, in addition to the support of recent peer reviewed literature illustrating a need for an appropriate criteria and more suitable speech recognition measure, believe it is appropriate at this time to re-evaluate the candidacy requirements associated with adult cochlear implantation. Specifically, this will be accomplished by evaluating the safety and efficacy of the Cochlear™ Nucleus® cochlear implant system under revised cochlear implant indications. The proposed approach would be to evaluate individuals scoring between 10 - 40% inclusively on Consonant Nucleus Consonant (CNC) monosyllabic words who do not meet current approved speech perception criteria with the widely used sentence measure Hearing In Noise Test (HINT) in quiet. No change to current qualifying audiometric criteria (bilateral moderate to profound sensorineural hearing loss in the low frequencies and profound hearing loss in the mid to high speech frequencies) for implant candidacy is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older at the time of the study.
* Preoperative aided CNC word score in quiet of greater than or equal to 10% and less than or equal to ¬¬40% in the ear to be implanted; equal to but no better than 50% in the contralateral ear
* Bilateral moderate to profound hearing loss in the low frequencies (up to 1000 Hz) and profound sensorineural hearing loss in the high speech frequencies (3000 Hz and above)
* Willingness to use bimodal stimulation (i.e. a cochlear implant on one ear and a hearing aid on the contralateral ear) through at least 6-months postactivation.
* English spoken as the primary language.

Exclusion Criteria:

* Congenital hearing loss (for the purpose of this study, onset prior to 2 years-of-age).
* Preoperative aided HINT sentence score less than or equal to 50% in the ear to be implanted
* Ossification, absence of cochlear development or any other cochlear anomaly that might prevent complete insertion of the electrode array.
* Hearing loss of neural or central origin (e.g., deafness due to lesions on the acoustic nerve or central auditory pathway).
* Active middle-ear infection.
* Unwillingness and/or inability of the candidate to comply with all investigational requirements including, but not limited to, study protocol and surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Driscoll, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Implanted: Subjects who met study inclusion and completed the primary endpoint of 6 months postimplant activation
Period: Overall Study
Arm/Group | Implanted
Started | 21 (subjects implanted)
Completed | 19 (subjects met the primary endpoint of 6 months postimplant activation)
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Subjects who met study inclusion and completed the primary endpoint of 6 months postimplant activation.
Arm/Group | Implanted
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 77 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Preoperative CNC word score - Treated Ear [Mean (Full Range); unit: percent correct] — Consonant Nucleus Consonant (CNC) Monosyllabic Word Test (Peterson & Lehiste, 1962). CNC Word Test is a validated test of open-set word recognition. The test consists of 10 lists with 50 monosyllabic words in each list. Subject responses are scored for words correct in the correct sequence. Subjects will be tested using a configuration of speech at 0º azimuth in quiet.
  percent correct | 23.6 [12 to 35]
Preoperative HINT Quiet score - Treated Ear [Mean (Full Range); unit: percent correct] — The Hearing in Noise Test (HINT) (Nilsson et al. 1994). The HINT sentences are recorded and consist of 25 equivalent lists. Each test list contains 10 sentences that vary from 3 to 7 words in length. Subjects will be tested in quiet using a configuration of speech at 0º azimuth in quiet.
  percent correct | 62.3 [47.2 to 86.4]
Preoperative AzBio Sentence Noise score - Treated Ear [Mean (Full Range); unit: percent correct] — AzBio Sentence Test (Spahr & Dorman, 2005). The AzBio Test is a validated test that consists of 15 lists of 20 sentences each. Each list includes 5 sentences from each of 4 different male and female speakers. Each word in the sentence counts towards the overall score. Subjects will be tested using a configuration of speech and noise at 0º azimuth.
  percent correct | 9.9 [0 to 34.8]

OUTCOME MEASURES:

1. Primary Outcome: CNC Monosyllabic Word Score - Treated Ear
Description: The primary study endpoint was to test whether a statistically significant difference could be obtained between the mean, preoperative Consonant Nucleus Consonant (CNC) monosyllabic word score in the ear to be implanted compared to the postoperative CNC word score in the cochlear implant alone condition at 6 months postimplant activation for candidates who currently perform outside the approved Nucleus® cochlear implant candidacy requirements.
  CNC Word Test is a validated test of open-set word recognition. The test consists of 10 lists with 50 monosyllabic words in each list. Subject responses are scored for both words and phonemes correct in the correct sequence. Subjects will be tested using a configuration of speech at 0º azimuth in quiet.
Time Frame: Six months
Measure: Mean (Full Range); unit: percent correct
Arm/Group | Implanted
Number analyzed (Participants) | 19
percent correct | 57.1 [16 to 95]

ADVERSE EVENTS:
Arm/Group | Implanted
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted (N=21)
Postoperative Pain (Ear and labyrinth disorders) | 1 — Postoperatively subject complained of local pain with reported questionable temperature. Antibiotics were prescribed as a precaution. One week following antibiotic course, no abnormalities were noted or reported.
Decrement in CNC word score performance postimplantation (Ear and labyrinth disorders) | 1 — Sentence testing: 37% pre-op, 36% 3 months, 53% 6 months. Subject stated memory affects performance. Integrity test results within normal limits (WNL) for receiver/stimulator and electrode array. Programming resolved sound quality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No